CLINICAL TRIAL: NCT05394636
Title: Cerebellar Superficial Siderosis in Cerebral Amyloid Angiopathy on 1.5T T2*-Weighted Imaging
Brief Title: Cerebellar Superficial Siderosis in Cerebral Amyloid Angiopathy
Acronym: CSS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/Dr-02
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Amyloid Angiopathy; Siderosis
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Siderosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cerebral amyloid angiopathy (CAA): Clinical and 1.5T MRI T2*-weighted imaging characteristics analyses from sporadic probable CAA patients (according to the modified Boston criteria) presenting with acute symptoms related to acute ICH, acute subarachnoid haemorrhage, or cortical SS,
  Interventions: Other: None, pure observational study

INTERVENTIONS:
Other: None, pure observational study — None, pure observational study

SUMMARY:
Cerebellar superficial siderosis (SS) has been recently reported to be present in about 10% of both hereditary (n=50) and sporadic (n=46) cerebral amyloid angiopathy (CAA) patients on 3T MRI using susceptibility-weighted imaging (SWI) in the majority of patients. In that study, cerebellar SS was associated with a higher number of supratentorial lobar and superficial cerebellar macrobleeds (although cerebellar SS was not directly located adjacent to these cerebellar macrobleeds). It is unclear if cerebellar SS is caused by in situ leakage of cerebellar leptomeningeal vessels or rather represents hemorrhagic diffusion from cerebellar parenchymal micro/macrobleeds or from supratentorial bleeding sources via the tentorium cerebelli (TC).

ELIGIBILITY:
Inclusion Criteria:

* CAA patients (according to the modified Boston criteria)
* with acute symptoms related to acute ICH, acute subarachnoid haemorrhage, or cortical SS

Exclusion Criteria:

* Patients with recent trauma,
* Patients with anticoagulation treatment,
* Patients with pathological blood coagulation tests (activated partial thromboplastin time [aPTT] ratio=patient's aPTT/normal control aPTT] >1.2; or partial thromboplastin time [PTT] <75%) or platelet count (<100 x 109/L)
* Patients with inflammatory CAA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sporadic probable CAA patients (according to the modified Boston criteria) presenting with acute symptoms related to acute ICH, acute subarachnoid haemorrhage, or cortical SS, between September 2009 and January 2022 in Nîmes University Hospital, France
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
MRI analyse : presence of cerebellar SS | baseline
  presence of cerebellar SS (Yes/No)
MRI analyse : Location of cerebellar SS | baseline
  Location of cerebellar SS (vermis, anterior lobe, posterior lobe)
MRI analyse : characteristics of cerebellar SS | baseline
  number of cerebellar sulci involved
MRI analyse : characteristics of cerebellar SS | baseline
  spatial relationship with cerebellar micro- and macrobleeds
MRI analyse : Presence of cerebellar macrobleeds | baseline
  Presence of cerebellar macrobleeds (Yes/No)
MRI analyse : Presence of cerebral macrobleeds | baseline
  Presence of cerebral macrobleeds (Yes/No)
MRI analyse : Characteristics of cerebral macrobleeds | baseline
  spatial relationship of cerebral macrobleeds with the TC [adjacent vs. non-adjacent to TC]
MRI analyse : Characteristics of cortical SS | baseline
  spatial relationship with TC (adjacent vs. non-adjacent to TC)
MRI analyse : hemosiderin | baseline
  presence of hemosiderin deposition along the TC.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Renard D, Laurent-Chabalier S, Leonte A, Hackius M, Parvu T, Wacongne A, Thouvenot E. Cerebellar Superficial Siderosis in Cerebral Amyloid Angiopathy on 1.5T T2*-Weighted Imaging. Cerebrovasc Dis. 2023;52(6):706-710. doi: 10.1159/000528384. Epub 2023 Mar 6. PMID 36878206